CLINICAL TRIAL: NCT03979027
Title: Acute Effects of Breakfast Compared With No Breakfast on Cognitive Function and Subjective State in 11-13 Year Old Children: A School-based, Randomised, Controlled, Parallel Groups Trial
Brief Title: Acute Effects of Breakfast Compared With No Breakfast on Cognitive Function and Subjective State in 11-13 Year Old Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Kellogg Company (Industry)
Responsible Party: Principal Investigator, Prof Louise Dye, Professor Louise Dye, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RTECCOG1113
Record Dates: First submitted 2019-06-03; First posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: Cognition
MeSH Terms: interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Breakfast (No Intervention): Fasting. Ad libitum water intake permitted.
- Breakfast (Experimental): Ad libitum intake of ready-to-eat-cereal with milk. Participants were given a choice of four commercially available RTECs with 1.8% fat cow's milk. Ad libitum water intake was also permitted. The four ready-to-eat-cereals were corn flakes, toasted rice, shredded whole wheat pieces with a sugar topping, and wheat, corn and oat shapes.
  Interventions: Dietary Supplement: Breakfast: ready-to-eat-cereal and milk

INTERVENTIONS:
Dietary Supplement: Breakfast: ready-to-eat-cereal and milk
  Arms: Breakfast

SUMMARY:
This study is a school-based, randomised, controlled, parallel groups trial to examine the acute effect of breakfast (ready-to-eat-cereal and milk) vs. no breakfast on cognitive function and subjective state in 11-13 year old adolescents. It was hypothesised that the consumption of breakfast will have a positive acute effect on cognitive performance and subjective state compared with breakfast omission in 11-13 year olds.

DETAILED DESCRIPTION:
This study is a school-based, randomised, controlled, parallel groups trial to examine the acute effect of breakfast (ready-to-eat-cereal and milk) vs. no breakfast on cognitive function and subjective state in 11-13 year old adolescents. It was hypothesised that the consumption of breakfast will have a positive acute effect on cognitive performance and subjective state compared with breakfast omission in 11-13 year olds. The study sample consisted of males and females aged 11-13 years who were recruited to take part in the study from a UK secondary school. There were two conditions in this parallel groups study: Breakfast and No breakfast (fasting). The breakfast intervention consisted of ad libitum intake of ready-to-eat-cereal with milk. Cognitive function was assessed at baseline and +70 and +215 minutes post-intervention. The Cambridge Neuro-psychological Test Automated Battery (CANTAB; Cambridge Cognition Ltd) was used to assess cognitive function. The battery included: Simple Reaction Time (SRT), 5-Choice Reaction Time (5-CRT), Rapid Visual Information Processing (RVIP), and Paired Associates Learning (PAL), which measured reaction time, visual-sustained attention, and visual-spatial memory respectively. Concomitant ratings of subjective mood, alertness, satiety, and motivation were taken throughout the morning using eight unipolar Visual Analogue Scales

ELIGIBILITY:
The inclusion criteria were as follows: aged 11-13 years, willingness to consume RTEC with semi-skimmed cow's milk during the study, ability to follow verbal and written instructions in English, and normal vision with appropriate corrective lenses if required. The exclusion criteria were as follows: inability to understand the objective of the cognitive tests or carry out the tests, behavioural difficulties or attention disorders, administration of any psychotropic medication in the month prior to testing or during testing, food allergies or intolerances which prevent consumption of RTEC and milk (e.g. coeliac, lactose intolerance), acute illness or feeling unwell within the week prior to testing or during testing, and hearing impairment that precluded the normal use of headphones.

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 234 (Actual)
Dates: Start 2011-01-04 (Actual); Primary Completion 2011-04-28 (Actual); Study Completion 2011-04-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline Paired Associates Learning (PAL) performance | baseline, 70 minutes post-intervention.
  Paired Associates Learning (PAL) task was administered on individual touchscreen portable computers.

SECONDARY OUTCOMES:
Simple Reaction Time task performance | baseline, 70 minutes and 215 minutes post-intervention
  Reaction time assessed by Simple Reaction Time (SRT) task. The task was administered on individual touchscreen portable computers.
5-Choice Reaction Time task performance | baseline, 70 minutes and 215 minutes post-intervention
  Reaction time assessed by 5-Choice Reaction Time (5-CRT) task. The task was administered on individual touchscreen portable computers.
Rapid Visual Information Processing task (RVIP) performance | baseline, 70 minutes and 215 minutes post-intervention
  Visual sustained attention assessed by Rapid Visual Information Processing task (RVIP). The task was administered on individual touchscreen portable computers.
Subjective unipolar visual analogue scale ratings of hunger | baseline, 15 minutes, 70 minutes, and 215 minutes post-intervention
  The unipolar Visual Analogue Scale is a horizontal line, 100mm in length, anchored by the extreme intensities of a single subjective feeling (e.g. 'not at all' to 'very'). The participant marks on the line at the point that they feel represents their perception of their current state. Participants responded to each Visual Analogue Scale using a touch screen computer by moving the cursor along a 100mm line with extreme anchors at each end. The initial location of the cursor was at the 50mm mark. There were 100 points on the scale, yielding possible scores of 0-100. Higher scores indicate a worse outcome
Subjective unipolar visual analogue scale ratings of cheerfulness | baseline, 15 minutes, 70 minutes, and 215 minutes post-intervention
  The unipolar Visual Analogue Scale is a horizontal line, 100mm in length, anchored by the extreme intensities of a single subjective feeling (e.g. 'not at all' to 'very'). The participant marks on the line at the point that they feel represents their perception of their current state. Participants responded to each Visual Analogue Scale using a touch screen computer by moving the cursor along a 100mm line with extreme anchors at each end. The initial location of the cursor was at the 50mm mark. There were 100 points on the scale, yielding possible scores of 0-100. Higher scores indicate a better outcome.
Subjective unipolar visual analogue scale ratings of energy | baseline, 15 minutes, 70 minutes, and 215 minutes post-intervention
  The unipolar Visual Analogue Scale is a horizontal line, 100mm in length, anchored by the extreme intensities of a single subjective feeling (e.g. 'not at all' to 'very'). The participant marks on the line at the point that they feel represents their perception of their current state. Participants responded to each Visual Analogue Scale using a touch screen computer by moving the cursor along a 100mm line with extreme anchors at each end. The initial location of the cursor was at the 50mm mark. There were 100 points on the scale, yielding possible scores of 0-100. Higher scores indicate a better outcome.
Subjective unipolar visual analogue scale ratings of motivation to try hard | baseline, 15 minutes, 70 minutes, and 215 minutes post-intervention
  The unipolar Visual Analogue Scale is a horizontal line, 100mm in length, anchored by the extreme intensities of a single subjective feeling (e.g. 'not at all' to 'very'). The participant marks on the line at the point that they feel represents their perception of their current state. Participants responded to each Visual Analogue Scale using a touch screen computer by moving the cursor along a 100mm line with extreme anchors at each end. The initial location of the cursor was at the 50mm mark. There were 100 points on the scale, yielding possible scores of 0-100. Higher scores indicate a better outcome
Subjective unipolar visual analogue scale ratings of ease of distraction | baseline, 15 minutes, 70 minutes, and 215 minutes post-intervention
  The unipolar Visual Analogue Scale is a horizontal line, 100mm in length, anchored by the extreme intensities of a single subjective feeling (e.g. 'not at all' to 'very'). The participant marks on the line at the point that they feel represents their perception of their current state. Participants responded to each Visual Analogue Scale using a touch screen computer by moving the cursor along a 100mm line with extreme anchors at each end. The initial location of the cursor was at the 50mm mark. There were 100 points on the scale, yielding possible scores of 0-100. Higher scores indicate a worse outcome
Subjective unipolar visual analogue scale ratings of ease of focusing | baseline, 15 minutes, 70 minutes, and 215 minutes post-intervention
  The unipolar Visual Analogue Scale is a horizontal line, 100mm in length, anchored by the extreme intensities of a single subjective feeling (e.g. 'not at all' to 'very'). The participant marks on the line at the point that they feel represents their perception of their current state. Participants responded to each Visual Analogue Scale using a touch screen computer by moving the cursor along a 100mm line with extreme anchors at each end. The initial location of the cursor was at the 50mm mark. There were 100 points on the scale, yielding possible scores of 0-100. Higher scores indicate a better outcome
Subjective unipolar visual analogue scale ratings of feeling of awake | baseline, 15 minutes, 70 minutes, and 215 minutes post-intervention
  The unipolar Visual Analogue Scale is a horizontal line, 100mm in length, anchored by the extreme intensities of a single subjective feeling (e.g. 'not at all' to 'very'). The participant marks on the line at the point that they feel represents their perception of their current state. Participants responded to each Visual Analogue Scale using a touch screen computer by moving the cursor along a 100mm line with extreme anchors at each end. The initial location of the cursor was at the 50mm mark. There were 100 points on the scale, yielding possible scores of 0-100. Higher scores indicate a better outcome
Subjective unipolar visual analogue scale ratings of bad temperedness | baseline, 15 minutes, 70 minutes, and 215 minutes post-intervention
  The unipolar Visual Analogue Scale is a horizontal line, 100mm in length, anchored by the extreme intensities of a single subjective feeling (e.g. 'not at all' to 'very'). The participant marks on the line at the point that they feel represents their perception of their current state. Participants responded to each Visual Analogue Scale using a touch screen computer by moving the cursor along a 100mm line with extreme anchors at each end. The initial location of the cursor was at the 50mm mark. There were 100 points on the scale, yielding possible scores of 0-100. Higher scores indicate a worse outcome
Subjective unipolar visual analogue scale ratings of cognitive test battery difficulty | baseline, 70 minutes, and 215 minutes post-intervention
  The unipolar Visual Analogue Scale is a horizontal line, 100mm in length, anchored by the extreme intensities of a single subjective feeling (e.g. 'not at all' to 'very'). The participant marks on the line at the point that they feel represents their perception of their cognitive test battery experience. Participants responded to each Visual Analogue Scale using a touch screen computer by moving the cursor along a 100mm line with extreme anchors at each end. The initial location of the cursor was at the 50mm mark. There were 100 points on the scale, yielding possible scores of 0-100. Higher scores indicate a worse outcome
Subjective unipolar visual analogue scale ratings of concentration during the cognitive test battery | baseline, 70 minutes, and 215 minutes post-intervention
  The unipolar Visual Analogue Scale is a horizontal line, 100mm in length, anchored by the extreme intensities of a single subjective feeling (e.g. 'not at all' to 'very'). The participant marks on the line at the point that they feel represents their perception of their cognitive test battery experience. Participants responded to each Visual Analogue Scale using a touch screen computer by moving the cursor along a 100mm line with extreme anchors at each end. The initial location of the cursor was at the 50mm mark. There were 100 points on the scale, yielding possible scores of 0-100. Higher scores indicate a better outcome
Subjective unipolar visual analogue scale ratings of performance on the cognitive test battery | baseline, 70 minutes, and 215 minutes post-intervention
  The unipolar Visual Analogue Scale is a horizontal line, 100mm in length, anchored by the extreme intensities of a single subjective feeling (e.g. 'not at all' to 'very'). The participant marks on the line at the point that they feel represents their perception of their cognitive test battery experience. Participants responded to each Visual Analogue Scale using a touch screen computer by moving the cursor along a 100mm line with extreme anchors at each end. The initial location of the cursor was at the 50mm mark. There were 100 points on the scale, yielding possible scores of 0-100. Higher scores indicate a better outcome
Subjective unipolar visual analogue scale ratings of frustration during the cognitive test battery | baseline, 70 minutes, and 215 minutes post-intervention
  The unipolar Visual Analogue Scale is a horizontal line, 100mm in length, anchored by the extreme intensities of a single subjective feeling (e.g. 'not at all' to 'very'). The participant marks on the line at the point that they feel represents their perception of their cognitive test battery experience. Participants responded to each Visual Analogue Scale using a touch screen computer by moving the cursor along a 100mm line with extreme anchors at each end. The initial location of the cursor was at the 50mm mark. There were 100 points on the scale, yielding possible scores of 0-100. Higher scores indicate a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Human Appetite Research Unit, University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adolphus K, Hoyland A, Walton J, Quadt F, Lawton CL, Dye L. Ready-to-eat cereal and milk for breakfast compared with no breakfast has a positive acute effect on cognitive function and subjective state in 11-13-year-olds: a school-based, randomised, controlled, parallel groups trial. Eur J Nutr. 2021 Sep;60(6):3325-3342. doi: 10.1007/s00394-021-02506-2. Epub 2021 Feb 20. PMID 33609174